CLINICAL TRIAL: NCT01435941
Title: Non-steroidal Anti-inflammatory Drugs Alone or With a Triptan and Reports of Transition From Episodic to Chronic Migraine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112630
Record Dates: First submitted 2011-09-08; First posted 2011-09-19 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Migraine Disorders
Keywords: mailed survey; non-steroidal anti-inflammatory drug; migraine disorders; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — Anti-Inflammatory Agents, Non-Steroidal; Tryptamines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Respondents who report episodic migraines (EM): Survey respondents whose headaches meet the diagnostic criteria for migraine and report that they experienced between 1 and 14 headache days in the month prior to the survey administration
  Interventions: Drug: Non-steroidal anti-inflammatory drug (NSAID); Drug: Triptan

INTERVENTIONS:
Drug: Non-steroidal anti-inflammatory drug (NSAID) — Participants who self-report that they have treated headaches with any drug in the non-steroidal anti-inflammatory drug (NSAID) class
Drug: Triptan — Participants who self-report that they have treated headaches with any drug in the NSAID class and any drug in the triptan class including naratriptan, sumatriptan, rizatriptan, frovatriptan, almotriptan, eletriptan, and zolmitriptan
  Other Names: Amerge® is a registered trademark of GlaxoSmithKline; Zomig® is a registered trademark of AstraZeneca; Relpax® is a registered trademark of Pfizer; Inc.; Maxalt® is a registered trademark of Merck & Co; Axert® is a registered trademark of Pharmacia; Frova® is a registered trademark of Elan Pharmaceuticals/UCB Pharma; Inc; Imitrex® is a registered trademark of GlaxoSmithKline

SUMMARY:
Chronic Migraine (CM), or 15 or more migraine headaches per month, is common in tertiary headache care and is associated with a number of deleterious outcomes, especially higher disability and poorer quality of life, relative to those with Episodic Migraine (EM) defined as 14 or fewer migraine headaches per month. Limited work has begun to examine factors that increase or decrease the risk of developing CM. One factor that appears especially relevant is symptomatic medication use. The current study builds upon and expands previous work considering the influence non-steroidal anti-inflammatory drug (NSAID) and/or triptan use has on the likelihood of developing CM.

This study is a retrospective observational cohort study of data collected via mail survey and collated in the American Migraine Prevalence and Prevention (AMPP) database.

Survey results from the AMPP study will be analyzed retrospectively. The AMPP is a longitudinal, population-based, mailed-questionnaire survey. In 2004, 120,000 United States (US) households were screened and 24,000 individuals who reported severe headaches were identified and additional questionnaires have been administered annually. This analysis uses data from respondents who meet second edition of the International Headache Classification-2 (IHCD-2) criteria for EM in 2005 with follow up results in 2006, 2007, 2008, and 2009. EM is defined as 1 to 14 headaches per month and CM is defined as 15 or more headaches per month.

ELIGIBILITY:
Inclusion Criteria:

* Respondents age 18 or older at the time of survey completion
* Respondents completed the questionnaires in 2004 and at least one other year (2005, 2006, 2007, 2008, 2009)
* Based on the respondents answers to the 2004 survey, their symptoms meet the criteria for EM which is characterized by headaches meeting International Classification of Headache Disorders - 2 (ICHD-2) criteria for migraine 1-14 days a month

Exclusion Criteria:

* Responses to questions suggest that the respondent's diagnosis is not migraine or CM

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The American Migraine Prevalence and Prevention (AMPP) study is a multi-year longitudinal population-based study that follows a cohort of headache sufferers with severe headaches. From 2004 to 2009, respondents with headaches completed mailed questionnaires. Respondents had been screened from 120,000 US households and 24,000 individuals with severe headaches were invited to respond to annual questionnaires. Within the 2005 EM cohort a transition was defined to have occurred if in the observed year a respondent was CM and in the year immediately preceding that year a subject was EM. Participants were followed for up to 4 years with the provision that the individual provided data in 2005 and then in at least one subsequent year (2006-2009).
Sampling Method: Non-Probability Sample
Enrollment: 11249 (Actual)
Dates: Start 2009-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of participants who progress from EM to CM | survey administered annually for 5 years
  The number of participants with episodic migraine (EM), characterized by headaches on 1 to 14 days per month, who report symptoms of chronic migraine (CM), 15 or more headaches per month, in one of the years of follow up

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline